CLINICAL TRIAL: NCT05483088
Title: Urine Sample Processing Study: Analysis of Fresh Versus Frozen Urine Samples From ICU Subjects
Brief Title: Urine Sample Processing Study
Status: Completed | Type: Observational
Sponsor: Astute Medical, Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: Turquoise
Record Dates: First submitted 2022-07-29; First posted 2022-08-01 (Actual); Last update posted 2023-10-26 (Actual); Status verified 2023-10

CONDITIONS: Acute Kidney Injury
MeSH Terms: conditions — Acute Kidney Injury | interventions — Urine Specimen Collection

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Urine
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes

GROUPS / COHORTS (1):
- Patients with KDIGO stage 2 or 3 AKI
  Interventions: Diagnostic Test: Urine collection for NEPHROCLEAR CCL14 Test

INTERVENTIONS:
Diagnostic Test: Urine collection for NEPHROCLEAR CCL14 Test — Urine will be collected for analysis with the NEPHROCLEAR CCL14 Test

SUMMARY:
The objective of the study is to collect and process urine samples from Intensive Care Unit (ICU) subjects with moderate to severe (Stage 2 or 3) acute kidney injury (AKI) for use in assessing the effects of urine sample freezing and various storage conditions on NEPHROCLEAR™ CCL14 Test results. This study is observational and will have no impact on the medical management of the subject.

ELIGIBILITY:
Inclusion Criteria:

1. Males and females 21 years of age or older;
2. Receiving care in an intensive care unit;
3. Expected to remain in the ICU for at least 48 hours after enrollment;
4. Use of indwelling urinary catheter as standard care at the time of enrollment;
5. Subject must have acute kidney injury (KDIGO Stage 2 or Stage 3) at the time of sample collection;
6. Urine sample must be collected within 36 hours of meeting KDIGO Stage 2 criteria;
7. Written informed consent provided by patient or legally authorized representative (LAR).

Exclusion Criteria:

1. Prior kidney transplantation;
2. Comfort-measures-only status;
3. Already receiving dialysis (either acute or chronic) or in imminent need of dialysis at the time of enrollment;
4. Known infection with human immunodeficiency virus (HIV) or active hepatitis (acute or chronic);
5. Special populations, pregnant women, prisoners or institutionalized individuals.

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult ICU patients with KDIGO stage 2 or 3 AKI.
Sampling Method: Non-Probability Sample
Enrollment: 110 (Actual)
Dates: Start 2021-11-12 (Actual); Primary Completion 2023-07-31 (Actual); Study Completion 2023-07-31 (Actual)

PRIMARY OUTCOMES:
Stability of CCL14 in urine samples | Up to 24 hours
  Stability of CCL14 in urine samples as measured by the NEPHROCLEAR™ CCL14 Test

CONTACTS AND LOCATIONS:
Locations (1):
- University of Maryland, Baltimore, Baltimore, Maryland, United States